CLINICAL TRIAL: NCT03916302
Title: Pulmonary Embolism WArsaw REgistry
Acronym: PE-aWARE
Status: Recruiting | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Piotr Pruszczyk, Prof., Medical University of Warsaw
Other Study IDs: PE-aWARE
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Acute Pulmonary Embolism
Keywords: acute pulmonary embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Complicated outcome: The patients meet at least one of the following criteria:
  1. systolic blood pressure < 90 mmHg for at least 15 minutes
  2. need for catecholamine administration because of persistant arterial hypotension or shock
  3. need for mechanical ventilation
  4. need for cardiopulmonary resuscitation
  5. bleeding classified according to the International Society on Thrombosis and Haemostasis classification (major bleeding and non-major clinically relevant bleeding).
- Non-complicated outcome: The patients meet none of the following criteria:
  1. systolic blood pressure < 90 mmHg for at least 15 minutes
  2. need for catecholamine administration because of persistant arterial hypotension or shock
  3. need for mechanical ventilation
  4. need for cardiopulmonary resuscitation
  5. bleeding classified according to the International Society on Thrombosis and Haemostasis classification (major bleeding and non-major clinically relevant bleeding).

SUMMARY:
Initiated in January 2008, The PE-aWARE (Pulmonary Embolism WArsaw REgistry) is an on-going single-centre prospective observational study of patients with confirmed acute pulmonary embolism (APE). Extensive data on consecutive patients with pulmonary embolism is collected and stored. The main objective is to collect and provide information on patients' characteristics, management, and outcome with the purpose of decreasing mortality in APE, the occurrence of bleeding, and the frequency of thromboembolic recurrences. Moreover, the PE-aWARE registry serves as a basis for creating predictive scores for clinicians which aid patient management. The study endpoints comprise clinically recognized (and objectively confirmed) recurrences of PE, major and minor bleeding complications classified according to the International Society on Thrombosis and Haemostasis classification, need for cardiopulmonary resuscitation or catecholamines, and death.

DETAILED DESCRIPTION:
The Pulmonary Embolism WArsaw REgistry (PE-aWARE) is an on-going prospective observational study of patients with confirmed acute pulmonary embolism (APE). Carried out since January 2008, the registry includes consecutive patients hospitalized at a single centre. The primary data recorded include details of each patient's clinical status, co-morbidities, the prescribed treatment, the results of additional studies (ie EKG, imaging studies), and the outcome. The study endpoints comprise clinically recognized (and objectively confirmed) recurrences of PE, major and minor bleeding complications classified according to the International Society on Thrombosis and Haemostasis classification, need for cardiopulmonary resuscitation or catecholamines, and death.

Collecting the fore mentioned data allows for clinicians to better manage the diagnostic workup and treatment and thus facilitates the prevention of possible future complications in APE patients.

ELIGIBILITY:
Inclusion Criteria:

* objectively confirmed pulmonary embolism
* Informed consent for the participation in the study, according to the requirements of the ethics committee

Exclusion Criteria:

* lack of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Concecutive patients hospitalized for pulmonary embolism
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2008-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite primary outcome | in-hospital (average of 10 days)
  at least one of the following:
  1. systolic blood pressure < 90 mmHg for at least 15 minutes
  2. need for catecholamine administration because of persistant arterial hypotension or shock
  3. need for mechanical ventilation
  4. need for cardiopulmonary resuscitation
Composite primary outcome | within 30 days from diagnosis
  at least one of the following:
  1. systolic blood pressure < 90 mmHg for at least 15 minutes
  2. need for catecholamine administration because of persistant arterial hypotension or shock
  3. need for mechanical ventilation
  4. need for cardiopulmonary resuscitation

SECONDARY OUTCOMES:
Major or non-major clinically relevant bleeding defined according to the International Society on Thrombosis and Haemostasis | in-hospital (average of 10 days)
  Secondary outcome measure
Major or non-major clinically relevant bleeding defined according to the International Society on Thrombosis and Haemostasis | within 30 days from diagnosis
  Secondary outcome measure

OTHER OUTCOMES:
5-year follow-up | 5 years
  Patients will be evaluated annually at least during first 5 years after index PE for VTE recurrence and for Post PE syndrome (PPS) including chronic thromboembolic pulmonary hypertension (CTEPH), chronic thromboembolic pulmonary disease (CTEPD), newly diagnosed neoplasms, cardiovascular diseases (coronary artery disease, stroke, heart failure) and functional limitation resulting from psychological sequel of acute PE.

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Pruszczyk, Prof., Study Director — Medical University of Warsaw
Locations (1):
- Department of Internal Medicine & Cardiology with the Centre for Management of Venous Thromboembolic Disease, Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No